CLINICAL TRIAL: NCT01011738
Title: A Multicenter, Prospective, Observational, Non-Interventional Cohort Study Evaluating On-Treatment Predictors of Response in Subjects With HBeAg Positive and HBeAg Negative Chronic Hepatitis B Receiving Therapy With PEGASYS(R) (Peginterferon Alfa-2a 40KD)
Brief Title: An Observational Cohort Study in Patients With Chronic Hepatitis B Receiving Pegasys
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MV22009
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational, non-interventional cohort study will evaluate predictors of response in patients with chronic hepatitis B receiving standard of care Pegasys therapy. Efficacy and safety parameters will also be evaluated. Patients included in the study will be followed for the duration of their treatment and for up to 3 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* adult patient, >/= 18 years of age
* chronic hepatitis B
* treatment with peginterferon alfa-2A

Exclusion Criteria:

* coinfection with HAV, HCV and HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C receiving treatment with peginterferon alfa-2a 40KD (Pegasys)
Sampling Method: Probability Sample
Enrollment: 1842 (Actual)
Dates: Start 2009-04-11 (Actual); Primary Completion 2014-11-18 (Actual); Study Completion 2014-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (249):
- Austria (5):
  - Lkh-Univ. Klinikum Graz, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Klinische Abt. Für Gaströnterologie & Hepatologie, Innsbruck
  - A.Ö. Krankenhaus Der Elisabethinen Linz; Iv. Med. Abtl., Linz
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin III - Gastroenterologie & Hepatologie, Vienna
  - Wilhelminenspital; Iv. Medizinische Abt., Vienna
- Salmaniya Medical Complex; Gastroenterology, Manama, Bahrain
- Bangladesh (2):
  - Liver Clinic Lab-Aid Specialized Hospital, Dhaka
  - The Liver Centre, Dhaka
- Bosnia and Herzegovina (7):
  - Clinical Center Banja Luka; Department for Infective Diseases, Banja Luka
  - Cantonal Hospital Bihac; Department for Infective Diseses, Bihać
  - Clinical Hospital Mostar; Department for Gastroenterology, Mostar
  - Clinical Center Sarajevo; Gastroenterohepatology, Sarajevo
  - University Clinical Center Tuzla; Clinic for Gastroenterology, Tuzla
  - University Clinical Center Tuzla; Clinic for Infective Diseases, Tuzla
  - Cantonal Hospital Zenica; Department for Infective Diseases, Zenica
- Bulgaria (2):
  - MHAT Tokuda Hospital Sofia; Department of Gastroenterology at Clinic of Internal Deseases, Sofia
  - Mhat Sveta Marina; Clinic of Gastroenterology, Varna
- China (23):
  - Beijing Ditan Hospital, Beijing
  - Beijing 302 Hospital; No. 2 Infectious Disease Section, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing You An Hospital; Digestive Dept, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital, Chongqing Medical University, Chongqing
  - The Eighth People's Hospital of Guangzhou, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Hangzhou Sixth People's Hospital, Hangzhou
  - The 1st Affiliated Hospital of Harbin Medical University, Harbin
  - Jinan Infectious Diseases Hospital, Jinan
  - Nanjing No.2 Hospital; Liver Disease Department, Nanjing
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - The 85th Hospital of P.L.A., Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Shenzhen Donghu Hospital, Shenzhen
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Bethune International Peace Hospital of PLA, Shijiazhuang
  - Xinjiang Uygur Autonomous Region Hospital of Chinese Traditional Medicine, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
- Egypt (8):
  - Gamal Sheha Clinic, Al Mansurah
  - Dr. Ibrahim Mostafa Clinic, Cairo
  - Yehia Elshazly Clinic for Hepatology and Gastroentrology, Cairo
  - Dr.Mohamed Amr Affifi Clinic, Cairo
  - Dr.Nabil Fawzy private clinic, Cairo
  - Dr.Nadia Elansary Clinic, Cairo
  - Dr. Taher Elzanaty clinic, Giza
  - Dr. Ahmed Monis Clinic, Giza
- France (65):
  - Ch Du Pays D Aix; Gastro Enterologie, Aix-en-Provence
  - Hopital Nord; Medecine A, Amiens
  - Hopital Nord; Reseau Hepatologie Picardie, Amiens
  - Hotel Dieu; Medecine A, Angers
  - Ch Victor Dupouy; Hepato Gastro Medecine Interne, Argenteuil
  - Ch Victor Dupouy; Oncologie, Argenteuil
  - Ch Henri Duffaut;Gastro Enterologie, Avignon
  - Hopital Jean Minjoz; Hepatologie, Besançon
  - Hopital Avicenne; Unite D Hepatologie, Bobigny
  - Hopital Jean Verdier; Gastro Enterologie, Bondy
  - Hopital Saint Andre; Hepato-Gastro-Enterologie, Bordeaux
  - Ch Pierre Oudot; Gastro Enterologie, Bourgoin
  - Hopital Cote De Nacre; Gastro Enterologie, Caen
  - Hopital Trousseau; Gastro Enterologie A Et B, Chambray-lès-Tours
  - Hopital Antoine Beclere; Hepatologie Gastro Enterologie, Clamart
  - Chu Estaing; Medecine Digestive, Clermont-Ferrand
  - Hopital Beaujon; Gastro Enterologie 1, Clichy
  - Hopital Beaujon;Hepatologie, Clichy
  - Ch Sud Francilien; Cons Gastro Enterologie, Corbeil-Essonnes
  - Ch Laennec; Medecine IV, Creil
  - Hopital Henri Mondor; Hepatologie Gastro Enterologie, Créteil
  - Hopital Du Bocage; Gastro Enterologie, Dijon
  - Ch Sud Francilien; Gastro Enterologie, Évry
  - CABINET, Grasse
  - Hopital Albert Michallon; Gastro Enterologie, La Tronche
  - Ch De Lagny Sur Marne; Gastro Enterologie, Lagny-sur-Marne
  - Ch De Bicetre; Gastro Enterologie, Le Kremlin-Bicêtre
  - Ch Du Mans; Medecine Ii, Le Mans
  - Hopital Claude Huriez;Gastro Enterologie, Lille
  - Hopital Dupuytren; Medecine Interne A, Limoges
  - Clinique De La Sauvegarde; Exploration Gastro Proctologie, Lyon
  - Hopital Hotel Dieu; Medecine Interne & D'Hepatologie, Lyon
  - Hopital De La Croix Rousse; Hepatologie Gastro Enterologie, Lyon
  - Fondation Hopital Saint Joseph; Gastro-Enterologie, Marseille
  - Hopital De La Conception; Gastro Enterologie Endoscopie 2E Nord, Marseille
  - Hopital De La Conception; Rhumatologie, Marseille
  - Hopital N D Bon Secours; Medecine B2, Metz
  - Ch De Montauban; Medecine Interne, Montauban
  - Hopital Jacques Monod; Gastro-Enterologie, Montivilliers
  - Cabinet Medical, Montpellier
  - Hopital Saint-Eloi; Hepatologie-Gastro-Enterologie, Montpellier
  - Hopital Emile Muller; Gastro Enterologie, Mulhouse
  - Hopital Hotel Dieu Et Hme; Hepatologie Gastro Enterologie, Nantes
  - Cabinet, Nantes
  - Ch Georges Renon; Maladies Infectieuses, Niort
  - Hopital Caremeau; Gastro Enterologie, Nîmes
  - Hopital La Source; Medecine H, Orléans
  - Fondation Institut Arthur Vernes; Institut Arthur Vernes, Paris
  - Hopital Saint Antoine; Hepatologie-Gastr-Enterologie, Paris
  - CH Pitie Salpetriere; Hepathologie Gastro Enterologie, Paris
  - Hopital Bichat Claude Bernard; Hepatologie Gastro Enterologie, Paris
  - Hopital Saint Jean; Hematologie, Perpignan
  - Hopital Du Haut-Leveque; Gastro-Enterologie, Pessac
  - Hopital Robert Debre; Gastro Enterologie, Reims
  - Hopital de Pontchaillou; Medicine Interne - Hepatologie, Rennes
  - Hopital Charles Nicolle; Gastro Enterologie, Rouen
  - Institut Arnault Tzanck; Medecine I Gastro Enterologie, Saint-Laurent-du-Var
  - Hopital Esquirol; Cons Externes, Saint-Maurice
  - Hopital Civil; Hepatologie-Gastro-Enterologie, Strasbourg
  - Cabinet Medical Gastro Enterologie, Toulon
  - Hopital Font Pre; Gastro Enterologie, Toulon
  - Hopital Purpan;Gastro Enterologie Hepatologie, Toulouse
  - Clinique Ambroise Pare; Medecine, Toulouse
  - Hopitaux de Brabois - Gastro-Entereologie, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse; Centre Hepatologie Biliaire, Villejuif
- Germany (37):
  - Charité Universitätsmedizin Berlin; Campus Mitte, Centrum 12, Medizinische Poliklinik, Berlin
  - Praxis Dr. med. Christine John, Berlin
  - überörtl.Gem.Praxis Dres. Stephan Dupke Axel Baumgarten, Berlin
  - Dres.Bernd Möller und Renate Heyne, Berlin
  - Praxis Dr. Heyne, Berlin
  - Charité - Campus Benjamin Franklin; Zentrum fuer Innere Medizin, Med. Klinik I, Berlin
  - Campus Virchow-Klinikum Charité Centrum 13; Medizinische Klinik; Abt.Hepatologie u.Gastroenterologie, Berlin
  - CAMPUS VIRCHOW-KLINIKUM; Charité Centrum 13; Med. Klinik Abt. Hepatologie u. Gastroenterologie, Berlin
  - Dres. Jörg Gölz und Arend Moll, Berlin
  - Universitätsklinikum Bonn Med. Klinik u. Poliklinik I, Bonn
  - Universitätsklinikum Klinik f. Gastroenterologie Hepatologie und Infektiologie, Düsseldorf
  - Universitätsklinikum Erlangen; Medizinische Klinik 1, Erlangen
  - Universitaetsklinikum Essen, Innere Klinik und Poliklinik fuer Tumorforschung, Essen
  - Praxis PD Dr.med. Gerlinde Teuber, Frankfurt am Main
  - Universitätsklinikum Freiburg Medizinische Klinik Innere Medizin I, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH Standort Gießen Medizinische Klinik II, Giessen
  - Med. Versorgungszentrum ifi-Institut, Hamburg
  - Infektionsmedizinisches Centrum Hamburg ICH Grindel, Hamburg
  - St.Marien-Hospital Klinik Knappenstraße Klinik f.Gastroenterologie, Hamm
  - Medizinische Hochschule Zentrum Innere Medizin Abt.Gastroenterologie, Endokrinologie und Hepatologie, Hanover
  - Uni Heidelberg Med. Klinik; Innere Medizin IV, Heidelberg
  - Dres.Dietrich Hüppe Gisela Felten und Heinz Hartmann, Herne
  - Universitätsklinikum Jena; Klinik für Innere Medizin II, Jena
  - Universitätsklinikum S.-H. Campus Kiel Klinik für Innere Medizin I Gastroenterologie Hepotologie, Kiel
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Med. Klinik I, Transplantationszentrum, Lübeck
  - Universitätsklinikum Magdeburg Klinik für Gastroenterologie und Hepatologie, Magdeburg
  - Uniklinik Mainz; I. Medizinische Klinik, Mainz
  - Klinikum rechts der Isar der TU München; II. Medizinische Klinik & Poliklinik, München
  - Dr.med.Heiner W.Busch und Stefan Christensen, Münster
  - Universitätsklinikum Münster Klinik und Poliklinik für Transplantationsmedizin, Münster
  - Klinikum Nord Medizinische Klinik 6, Nuremberg
  - St. Josefs Klinik; Medizinische Klinik, Offenburg
  - Klinikum Salzgitter-Lebenstedt Medizinische Klinik I, Salzgitter
  - Dres. Andreas Schaffert Andreas Trein und Edith Ißler u.w., Stuttgart
  - Universitätsklinikum Ulm; Medizinische Uni-Klinik III Abt. Innere Medizin III Hämatologie u. Onkolo., Ulm
  - Praxis Sabine Mauruschat, Wuppertal
  - Medizinische Universitätsklinik; Med. Klinik Ii, Infektiologie, Würzburg
- Tuen Mun Hospital; Medicine & Geriatrics, Tuenmen, Hong Kong
- India (8):
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Institute of Digestive Diseases, Guwahati
  - Medanta -The Medicity; Department of Digestive and Hepatobiliary Sciences, Gūrgaon
  - Opp Jaslok Hospital, Mumbai
  - Krishnai Clinic, Pune
  - Medipoint Clinic, Pune
  - Pai Clinic and Diagnostic Center, Pune
  - Sree Gokulam Medical College and Research Foundation, Trivandrum
- Indonesia (12):
  - Boromeus Hospital; Hepatology, Bandung
  - Santosa Bandung International Hospital; Hepatology, Bandung
  - Hasan Sadikin Hospital; Digestive Surgery, Bandung
  - Klinik Hati; Hepatology, Jakarta
  - PGI Cikini Hospital; Hepatology, Jakarta
  - Central Army Hospital Rspad Gatot Soebroto; Pulmonology, Jakarta
  - Cipto Mangunkusumo General Hospital; Hematology & Oncology, Jakarta
  - Medistra Hospital; Hepatology, Jakarta
  - Mitra International Jatinegara Hospital; Hepatology, Jakarta
  - Klinik Kimia Farma, Jakarta
  - Dr. Soetomo Hospital; Kidney and Hipertansion, Surabaya
  - Bintaro International Hospital, Hepatology, Tangerang
- Ireland (2):
  - Mater Misericordiae University Hospital;Gastrointestinal Unit/Center for Liver Disease, Dublin
  - St. James Hospital; Hepatology, Dublin
- Jordan (3):
  - Al-Bashir Hospital, Amman
  - Prince Hamzeh Hospital; Internal Medicine, Amman
  - King Abdullah University Hospital, Irbid
- Lebanon (3):
  - American University of Beirut - Medical Center, Beirut
  - Beirut Governmental University Hospital, Beirut
  - Hotel-Dieu de France Hospital; Gastroenterology, Beirut
- Morocco (3):
  - Cabinet Privé Pr D Jamil, Casablanca
  - CHU Hassan 2; Service Gastro Enterologie Pr IBRAHIMI, Fes
  - Centre Hospitalier Universitaire Ibn Sina; Service de Gastro-entérologie Essaid, Rabat
- New Zealand (3):
  - Auckland Hospital; New Zealand Liver Transplant Unit, Auckland
  - Waikato Hospital; Gastroenterology, Hamilton
  - Hepatitis Foundation, Whakatane
- North Macedonia (2):
  - Clinical Center Skopje; Gastroenterohepatology, Skopje
  - Clinical Center Skopje; Infectious Diseases, Skopje
- Pakistan (10):
  - Allied Hospital; Department of Medicine, Faisalabad
  - Islamabad Specialist Clinic, Islamabad
  - Akbar Center, Karachi
  - Dow University of Health Sciences; Department of Medicine, Karachi
  - Medicare Clinics, Karachi
  - Sheikh Zayed Hospital; Department of Gastroentrology, Lahore
  - Kanaan Clinic, Lahore
  - Saeed Anwar Medical Centre, Peshawar
  - Combined Military Hospital; Department of Medicine, Rawalpindi
  - Holy Family Hospital; Department of Medicine, Rawalpindi
- Poland (13):
  - Medical Uni of Bialystok; Infectious Diseases, Bialystok
  - Hospital For Infectious Diseases; Infectiology, Bydgoszcz
  - Szpital Specjalistyczny; Oddzial Obserwacyjno - Zakayny, Chorzów
  - Pomorskie Centrum Chorob Zakaznych i Gruzlicy, Gdansk
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II; Oddzial Wirusowego Zapalenia Watroby, Krakow
  - Medical Uni of Lodz; Infectious Diseases, Lodz
  - Specjalistyczny Szpital Wojewódzki im. Biegańskiego; Klinika Chorób Zakaźnych i Hepatologii UM, Lodz
  - Wojewódzki specjalistyczny szpital im. Bieganskiego; Oddział Obserwacyjno-Zakazny i Chorob Watroby, Lodz
  - Inst. of Infectious & Parasitic Diseases; Clinic of Hepatology & Aquired Immunodeficiencies, Warsaw
  - Centralny Szpital Kliniczny MSWiA; Oddzial Chorob Wewnetrznych i Hepatologii, Warsaw
  - Wojewodzki Szpital; Specjalistyczny Chorob Zakaznych, Wroclaw
  - NZOZ Lubuska Specjalistyczna Poradnia Chorob Watroby, Zielona Góra
  - Centrum Medyczne, Łańcut
- Portugal (3):
  - Hospital de Santa Maria; Servico de Gastrenterologia e Hepatologia, Lisbon
  - Hospital Geral de Santo Antonio; Servico de Gastrenterologia, Porto
  - Hospital de Sao Joao; Servico de Gastrenterologia, Porto
- Romania (5):
  - Cantacuzino Clinical Hospital;Gastroenterology Department, Bucharest
  - Institutul De Boli Infectioase Matei Bals; Sectia Clinica II Boli Infectioase Adulti, Bucharest
  - The Hospital of Tropical and Infectious Disease Victor Babes, Bucharest
  - Clinical Infectious Diseases Hospital Victor Babes, Craiova
  - Spitalul Clinic de Boli Infectioase si Tropicale Dr. Victor; INFECTIOUS DISEASE, Craiova
- Saudi Arabia (5):
  - King Fahad University Hospital; Internal Medicine, Khobar
  - Riyadh Military Hospital, Riyadh
  - King Faisal Specialist Hospital & Research Centre; Oncology, Riyadh
  - King Fahad Medical City; Gastroentrology, Riyadh
  - North West Armed Forces Hospital; Internal Medicine, Tabuk
- South Korea (15):
  - Pyungchon Sacred Heart Hospital, Anyang
  - Pusan University Hospital, Busan
  - Inje University Pusan Paik Hospital, Busan
  - Chooncheon Sacred Heart Hospital, Chooncheon
  - Kyungpook National Uni Hospital; Internal Medicine, Daegu
  - Chungnam University Hospital, Daejeon
  - Inha University Hospital, Incheon
  - Chonbuk National Uni Hospital, Jeollabuk-do
  - Eulji General Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - Yonsei Uni College of Medicine, Severance Hospital; Internal Medicine Dept., Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - Korea Kuro Hospital; Internal Medicine, Seoul
  - Pundang Jesaeng General Hospital, Seoungnamsi
  - Ulsan University Hosiptal, Ulsan
- Thailand (3):
  - Siriraj Hospital, Bangkok
  - Chiang Mai Uni Hospital; Faculty of Medicine, Chiang Mai
  - Songklanagarind Hospital; Division of Gastroenterology, Songkhla
- Rashid Hospital; Gastroenterology, Dubai, United Arab Emirates
- United Kingdom (7):
  - Hull Royal Infirmary; Department Hepatology and Gastroenterology, Hull
  - The Royal London Hospital, London
  - King'S College Hospital, London
  - St. Georges Uni of London; Gastroenterology & Hepatology, London
  - University College London; Hepatology, London
  - Imperial College Healthcare Trust, London
  - Manchester Royal Infirmary; Department Of Medicine, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1842 participants were enrolled at 219 centers across 26 countries from 10 April 2009 to 17 November 2014.
Groups:
- HBeAg Positive: This group included participants who tested positive for Hepatitis B envelope antigen (HBeAg) when entering the study. Hepatitis B envelope antigen is a protein from the Hepatitis B virus that circulates in infected blood when the virus is actively replicating. The presence of HBeAg suggests that the participant is infectious and is able to spread the virus to other people.
- HBeAg Negative: This group included participants who tested negative for Hepatitis B envelope antigen (HBeAg) when entering the study. HBeAg-negative Hepatitis B is a form of the virus that does not cause infected cells to secrete HBeAg. Participant can be infected with the HBeAg-negative form of the virus from the beginning, or the viral mutation can emerge later in the course of infection in participant initially infected with the HBeAg-positive form of the virus. HBeAg-negative chronic hepatitis is thus characterized by detection of HBsAg without HBeAg in serum.
- HBeAg Status Unknown: This group included participants with Chronic Hepatitis B (CHB) virus infection whose HBeAg status was not known.
Period: Overall Study
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown
Started | 877 | 912 | 53
Completed | 553 | 618 | 36
Not Completed | 324 | 294 | 17
Not completed — Death | 12 | 3 | 0
Not completed — Unknown reasons | 312 | 291 | 17

BASELINE CHARACTERISTICS:
Population: Safety population was defined to include participants with informed consent who received at least one dose of peginterferon alfa-2a and had at least one post-baseline safety assessment (any assessment after baseline).
Groups:
- Total: Total of all reporting groups
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown | Total
Number analyzed (Participants) | 863 | 890 | 48 | 1801
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (9.37) | 37.8 (10.81) | 38.6 (12.69) | 34.6 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257 | 231 | 11 | 499
  Male | 606 | 659 | 37 | 1302

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus Surface Antigen Clearance
Description: Percentage of participants who became Hepatitis B Virus Surface Antigen (HBsAg) negative by the end of the observation period. A participant was considered to have achieved HBsAg clearance if the HBsAg measurement was reported as: (a) 'Negative' or (b) a quantitative result lower than the reported lower limit of detection. An observational period was upto 3 years post-treatment. The analysis was performed by 2 methods: Analysis A and Analysis B. For analysis A, all participants included in the analyzed population were used (participants with missing measurement for calculation of the endpoint were considered non-responders regarding the endpoint). For analysis B method, only participants in the analyzed population without missing measurements for calculation of the endpoint were used (analysis "as observed").
Time Frame: Up to 276 Weeks
Population: mITT population included all participants of the target population who could be classified regarding their HBeAg status. The target analysis population was per the inclusion/exclusion criteria mentioned in the protocol. Data of participants available at the assessment time point were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Percentage of Participants
  Analysis A, n= 844, 872 | 2 [1 to 3] | 5 [3 to 6]
  Analysis B, n= 328, 394 | 5 [3 to 8] | 10 [8 to 14]

2. Secondary Outcome: Percentage of Participants With Suppression of Hepatitis B Virus Deoxyribonucleic Acid to <2,000 International Units Per Milliliter
Description: A participant was considered to have achieved suppression of Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) to <2,000 International Units Per Milliliter (IU/mL) if the HBV DNA measurement is lower than 2,000 IU/mL.
Time Frame: Up to 276 Weeks
Population: mITT population included all participants of the target population who could be classified regarding their HBeAg status. The target analysis population was per the inclusion/exclusion criteria mentioned in the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Percentage of Participants
  End of treatment, Analysis A, n= 844, 872 | 39 [36 to 43] | 70 [67 to 73]
  End of treatment, Analysis B, n= 616,612 | 54 [50 to 58] | 89 [86 to 91]
  6 months post-treatment, Analysis A, n= 844, 872 | 24 [21 to 27] | 33 [30 to 36]
  6 months post-treatment, Analysis B, n= 584, 634 | 34 [31 to 38] | 45 [41 to 49]
  1 year post-treatment, Analysis A, n = 844, 872 | 20 [17 to 23] | 23 [20 to 26]
  1 year post-treatment, Analysis B, n = 525,557 | 32 [28 to 37] | 36 [32 to 40]
  2 year post-treatment, Analysis A, n = 844, 872 | 18 [15 to 21] | 19 [16 to 21]
  2 year post-treatment, Analysis B, n = 505, 534 | 30 [26 to 34] | 30 [26 to 34]
  3 year post-treatment, Analysis A, n = 844, 872 | 13 [11 to 16] | 16 [14 to 19]
  3 year post-treatment, Analysis B, n = 421,448 | 27 [23 to 31] | 31 [27 to 36]

3. Primary Outcome: Predictive Values of Early on Treatment Response for Hepatitis B Surface Antigen Clearance 3 Years Post-Treatment- Hepatitis B Virus e Antigen Positive Participants
Description: The probability that the participant who develops an early virological/serological response would achieve Hepatitis B Surface Antigen (HBsAg) clearance 3 years post-treatment is called the positive predictive value (PPV) of the early virological/serological response. The probability that the participant who fails to develop an early virological/serological response also would fail to achieve HBsAg clearance 3 years post-treatment is called the negative predictive value (NPV) of the early virological/serological response. The positive and negative predictive values of early response at Weeks 12 and 24 on achievement of HBsAg clearance at 3 years post-treatment were examined. The following evidence of early response was explored (giving both NPV and PPV): For HBeAg positive participant, HBsAg <1,500 International Units Per Milliliter (IU/mL) and HBsAg <20,000 IU/mL at Weeks 12 and 24.
Time Frame: Up to 276 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive
Number analyzed (Participants) | 844
Percentage of Participants
  HBsAg<1500 IU/mL at Week 12, n=410,PPV, Analysis A | 4 [1 to 11]
  HBsAg<1500 IU/mL at Week 12, n=171,PPV, Analysis B | 11 [3 to 27]
  HBsAg<1500 IU/mL at Week 12, n=410,NPV, Analysis A | 99 [97 to 100]
  HBsAg<1500 IU/mL at Week 12, n=171,NPV, Analysis B | 98 [94 to 100]
  HBsAg<20000 IU/mL at Week 12, n=410,PPV,Analysis A | 2 [1 to 4]
  HBsAg<20000 IU/mL at Week 12, n=171,PPV,Analysis B | 4 [1 to 9]
  HBsAg<20000 IU/mL at Week 12, n=410,NPV,Analysis A | 98 [93 to 100]
  HBsAg<20000 IU/mL at Week 12, n=171,NPV,Analysis B | 95 [84 to 99]
  HBsAg<1500 IU/mL at Week 24, n=374,PPV, Analysis A | 5 [2 to 11]
  HBsAg<1500 IU/mL at Week 24, n=167,PPV, Analysis B | 11 [4 to 22]
  HBsAg<1500 IU/mL at Week 24, n=374,NPV, Analysis A | 99 [97 to 100]
  HBsAg<1500 IU/mL at Week 24, n=167,NPV, Analysis B | 98 [94 to 100]
  HBsAg<20000 IU/mL at Week 24,n=374, PPV,Analysis A | 2 [1 to 5]
  HBsAg<20000 IU/mL at Week 24, n=167,PPV,Analysis B | 5 [2 to 11]
  HBsAg<20000 IU/mL at Week 24,n=374, NPV,Analysis A | 99 [94 to 100]
  HBsAg<20000 IU/mL at Week 24, n=167,NPV,Analysis B | 97 [85 to 100]
Statistical Analysis 1: Comparison: HBeAg Positive; In HBeAg positive participants, Log10-drop HBsAg at Week 24 was analyzed as the predictor factor of HBsAg clearance at 3 years post-treatment in analysis A; Test type: Superiority or Other; p = 0.0022, Wald-Chi-Square test — Multiple logistic regression were run in stepwise procedure with significance level of 0.05 to stay, considering all pre and on-treatment factors identified by univariate logistic regression to be associated with HBsAg clearance 3 yrs post-treatment; Odds Ratio (OR) = 3.349, 95% CI 2-sided [1.542 to 7.271]
Statistical Analysis 2: Comparison: HBeAg Positive; In HBeAg positive participants, Log10-drop HBsAg at Week 24 was analyzed as the predictor factor of HBsAg clearance at 3 years post-treatment in analysis B; Test type: Superiority or Other; p = 0.0019, Wald-Chi-Square test — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.595, 95% CI 2-sided [1.603 to 8.063]
Statistical Analysis 3: Comparison: HBeAg Positive; In HBeAg positive participants, Weight in kg was analyzed as independent predictor factor of HBsAg clearance at 3 years post-treatment in analysis A; Test type: Superiority or Other; p = 0.0369, Wald-Chi-Square test — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.851, 95% CI 2-sided [0.732 to 0.990]

4. Secondary Outcome: Percentage of Participants With Hepatitis B Virus e Antigen Seroconversion in Hepatitis B Virus e Antigen Positive Participants
Description: HBeAg seroconversion is presented as percentage of participants who become HBeAg negative and anti-HBe positive. A participant was considered to have achieved HBeAg seroconversion if (a) the participant achieved HBeAg loss and (b) the anti-HBe measurement was reported as (i) 'POSITIVE' or (ii) a quantitative result considered 'positive' in the context. HBeAg seroconversion and suppression of HBV DNA to <2,000 IU/mL: A participant was considered to have achieved HBeAg seroconversion and suppression of HBV DNA to <2,000 IU/mL if (a) the participant achieved HBeAg seroconversion and (b) the participant achieved suppression of HBV DNA to <2,000 IU/mL.
  Abbreviations for pt=post-treatment.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive
Number analyzed (Participants) | 844
Percentage of Participants
  EOT, HBeAg seroconversion, n=844,Analysis A | 14 [11 to 16]
  EOT, HBeAg seroconversion, n=509,Analysis B | 23 [19 to 27]
  6 months pt,HBeAg seroconversion, n=844,Analysis A | 16 [14 to 19]
  6 months pt,HBeAg seroconversion, n=486,Analysis B | 28 [24 to 32]
  1 yr pt, HBeAg seroconversion, n=844, Analysis A | 17 [14 to 19]
  1 yr pt, HBeAg seroconversion, n=438, Analysis B | 32 [28 to 37]
  2 Yrs pt,HBeAg seroconversion, n=844,Analysis A | 18 [16 to 21]
  2 Yrs pt,HBeAg seroconversion, n=398, Analysis B | 39 [34 to 44]
  3 Yrs pt,HBeAg seroconversion, n=844, Analysis A | 14 [11 to 16]
  3 Yrs pt,HBeAg seroconversion, n=304, Analysis B | 38 [32 to 44]

5. Secondary Outcome: Percentage of Participants With Hepatitis B Virus e Antigen Loss in Hepatitis B Virus e Antigen Positive Participants
Description: A participant was considered to have achieved HBeAg loss if the HBeAg measurement was reported as (a) 'NEGATIVE' or (b) a quantitative result was lower than the reported lower detection limit. This endpoint was measured in the participants with HBeAg positive CHB.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive
Number analyzed (Participants) | 844
Percentage of Participants
  EOT, HBeAg loss, n=844, Analysis A | 18 [15 to 20]
  EOT, HBeAg loss, n=554, Analysis B | 27 [23 to 31]
  6 months pt, HBeAg loss, n=844, Analysis A | 21 [19 to 24]
  6 months pt, HBeAg loss, n=516, Analysis B | 35 [31 to 39]
  1 yr pt, HBeAg loss, n=844, Analysis A | 22 [19 to 24]
  1 yr pt, HBeAg loss, n=460, Analysis B | 40 [35 to 44]
  2 yr pt, HBeAg loss, n=844, Analysis A | 23 [21 to 26]
  2 yr pt, HBeAg loss, n=430, Analysis B | 46 [41 to 51]
  3 yr pt, HBeAg loss, n=844, Analysis A | 19 [17 to 22]
  3 yr pt, HBeAg loss, n=331, Analysis B | 49 [44 to 55]

6. Secondary Outcome: Percentage of Participants With Hepatitis B Virus e Antigen Seroconversion and Hepatitis B Virus Deoxyribonucleic Acid <2000IU/mL in Hepatitis B Virus e Antigen Positive Participants
Description: A participant was considered to have achieved HBeAg seroconversion and suppression of HBV DNA to <2,000 IU/mL if (a) the participant achieved HBeAg seroconversion and (b) the participant achieved suppression of HBV DNA to <2,000 IU/mL. If a patient received NUCs after end of PEG IFN treatment, then a reported suppression of HBV DNA to < 2,000 IU/mL during or after this NUC treatment were to be ignored, and HBV DNA ≥ 2,000 IU/mL was to be assigned. However, HBV DNA < 2,000 IU/mL was not to be ignored, if the NUC treatment given parallel to PEG IFN was discontinued within the first 8 weeks after end of PEG IFN treatment and prior to the HBV DNA value concerned no further NUCs were administered.
  Abbreviations for Seroconversion=sercnvrsn, Analysis A= AnalysA, and Analysis B= AnalysB, pt=post-treatment.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive
Number analyzed (Participants) | 844
Percentage of Participants
  EOT,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=844,AnalysA | 11 [9 to 14]
  EOT,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=480,AnalysB | 20 [17 to 24]
  6 m,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=844,AnalysA | 9 [8 to 12]
  6 m,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=461,AnalysB | 17 [14 to 21]
  1yr,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=844,AnalysA | 7 [5 to 9]
  1yr,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=415,AnalysB | 14 [11 to 18]
  2yr,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=844,AnalysA | 7 [5 to 9]
  2yr,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=383,AnalysB | 16 [12 to 20]
  3yr,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=844,AnalysA | 5 [4 to 7]
  3yr,HBeAg sercnvrsn/HBVDNA<2000IU/mL,n=285,AnalysB | 15 [11 to 20]

7. Primary Outcome: Predictive Values of Early on Treatment Response for Hepatitis B Surface Antigen Clearance 3 Years Post-Treatment- Hepatitis B Virus e Antigen Negative Participants
Description: The probability that the participant who develops an early virological/serological response would achieve HBsAg clearance 3 years post-treatment is called the PPV of the early virological/serological response. The probability that the participant who fails to develop an early virological/serological response also would fail to achieve HBsAg clearance 3 years post-treatment is called the NPV of the early virological/serological response. The positive and negative predictive values of early response at Weeks 12 and 24 on achievement of HBsAg clearance at 3 years post-treatment were examined. The following evidence of early response was explored (giving both NPV and PPV): For HBeAg negative patients, any decline in HBsAg from baseline to Week 12 and 24 and at least a 10% decline in HBsAg from baseline to Weeks 12 and 24.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Negative
Number analyzed (Participants) | 872
Percentage of Participants
  Any HBsAg decline to Week 12,n=310, PPV,Analysis A | 7 [4 to 12]
  Any HBsAg decline to Week 12,n=161,PPV, Analysis B | 13 [7 to 22]
  Any HBsAg decline to Week 12,n=310, NPV,Analysis A | 98 [94 to 100]
  Any HBsAg decline to Week 12,n=161,NPV, Analysis B | 96 [88 to 99]
  HBsAg decline>=10% to Week 12,n=310,PPV,Analysis A | 8 [4 to 14]
  HBsAg decline>=10% to Week 12,n=161,PPV,Analysis B | 16 [8 to 26]
  HBsAg decline>=10% to Week 12,n=310,NPV,Analysis A | 98 [95 to 100]
  HBsAg decline>=10% to Week 12,n=161,NPV,Analysis B | 96 [90 to 99]
  Any HBsAg decline to Week 24,n=286, PPV,Analysis A | 7 [4 to 12]
  Any HBsAg decline to Week 24,n=147,PPV,Analysis B | 15 [8 to 24]
  Any HBsAg decline to Week 24,n=286, NPV,Analysis A | 99 [94 to 100]
  Any HBsAg decline to Week 24,n=147,NPV,Analysis B | 98 [90 to 100]
  HBsAg decline>=10% to Week 24,n=286,PPV,Analysis A | 8 [4 to 13]
  HBsAg decline>=10% to Week 24,n=147,PPV,Analysis B | 17 [10 to 27]
  HBsAg decline>=10% to Week 24,n=286,NPV,Analysis A | 99 [95 to 100]
  HBsAg decline>=10% to Week 24,n=147,NPV,Analysis B | 98 [92 to 100]
Statistical Analysis 1: Comparison: HBeAg Negative; In HBeAg negative participants, HBsAg in log10 IU/mL at Week 24 was analyzed as the predictor factor of HBsAg clearance at 3 years post-treatment in analysis A; Test type: Superiority or Other; p = 0.0033, Wald-Chi-Square test — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.155, 95% CI 2-sided [0.045 to 0.539]
Statistical Analysis 2: Comparison: HBeAg Negative; In HBeAg negative participants, HBsAg in log10 IU/mL at Week 24 was analyzed as the predictor factor of HBsAg clearance at 3 years post-treatment in analysis B; Test type: Superiority or Other; p = 0.0042, Wald-Chi-Square test; Odds Ratio (OR) = 0.191, 95% CI 2-sided [0.062 to 0.594]
Statistical Analysis 3: Comparison: HBeAg Negative; In HBeAg negative participants, ALT ratio was analysed as the predictor factor of HBsAg clearance at 3 years post-treatment in analysis A; Test type: Superiority or Other; p = 0.0149, Wald-Chi-Square test — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.528, 95% CI 2-sided [1.086 to 2.150]

8. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen Seroconversion
Description: Hepatitis B surface antigen (HBsAg) is a viral protein detectable in the blood in acute and chronic hepatitis B infection. A participant was considered to have achieved HBsAg seroconversion if (a) the participant achieved HBsAg clearance and (b) the last approved anti-HBs measurement in the analyzed time window was reported as i) 'POSITIVE' or (ii) quantitative result and was greater than or equal to the reported lower limit of detection.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Percentage of Participants
  EOT, n=844,872, Analysis A | 2 [1 to 3] | 1 [1 to 3]
  EOT, n=338,286, Analysis B | 5 [3 to 8] | 5 [2 to 8]
  6 months post-treatment, n=844,872, Analysis A | 2 [1 to 3] | 3 [2 to 4]
  6 months post-treatment, n=318,254, Analysis B | 5 [3 to 8] | 9 [6 to 14]
  1 Year post-treatment, n=844,872, Analysis A | 2 [1 to 3] | 2 [1 to 3]
  1 Year post-treatment, n=285,239, Analysis B | 6 [4 to 10] | 8 [5 to 12]
  2 Year post-treatment, n=844,872, Analysis A | 2 [1 to 3] | 1 [1 to 2]
  2 Year post-treatment, n=257,217, Analysis B | 5 [3 to 9] | 5 [3 to 9]
  3 Year post-treatment, n=844,872, Analysis A | 1 [0 to 2] | 2 [1 to 3]
  3 Year post-treatment, n=193,179, Analysis B | 5 [2 to 9] | 9 [5 to 14]

9. Secondary Outcome: Quantitative Hepatitis B Surface Antigen
Description: Quantitative HBsAg assay is a diagnostic test for assessing the amount of the HBsAg in chronic hepatitis B participants. Last approved quantitative HBsAg measurement in the analyzed time window.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Log10 IU/mL
  Baseline, HBsAg in log10 IU/mL, n=354, 370 | 3.94 (0.76) | 3.45 (0.84)
  Decline at Week 12 in log10 IU/mL,n=286,210 | 0.32 (0.69) | 0.18 (0.61)
  Decline at Week 24 in log10 IU/mL, n=251,286 | 0.57 (1.01) | 0.39 (0.81)
  Decline at Week 36 in log10 IU/mL, n=149, 182 | 0.79 (1.18) | 0.44 (0.81)
  Decline at week 48 in log10 IU/mL, n=161,240 | 0.99 (1.34) | 0.60 (0.97)
  Decline at end of trt. in log10 IU/mL, n=233,278 | 0.79 (1.27) | 0.56 (0.95)
  Decline 6 month pt. in log10 IU/mL, n=190,242 | 0.76 (1.24) | 0.54 (0.93)
  Decline 1 year pt. in log10 IU/mL, n=142,180 | 0.79 (1.31) | 0.58 (1.07)
  Decline 2 years pt. in log10 IU/mL, n=132,137 | 0.90 (1.29) | 0.56 (0.98)
  Decline 3 years pt. in log10 IU/mL, n=104, 126 | 0.82 (1.18) | 0.75 (1.02)

10. Secondary Outcome: Percentage of Participants With Normalization of Alanine Transaminase
Description: A participant was considered to have achieved normalization of alanine transaminase (ALT) if the ALT measurement was lower or equal to the upper limit of the normal range. Only patients with elevated ALT at baseline were included in any analyses where normalization of ALT was used as endpoint. It was analyzed as last serum ALT in the analyzed time window, divided by the upper limit of the normal range.
Time Frame: Up to 276 Weeks
Population: mITT included all participants of the target population who could be classified regarding their HBeAg status. The target analysis population was per the inclusion/exclusion criteria mentioned in the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 751 | 610
Percentage of Participants
  Week 12, n=751,610, Analysis A | 23 [20 to 26] | 23 [20 to 26]
  Week 12, n=685,564, Analysis B | 25 [22 to 29] | 25 [21 to 28]
  Week 24, n=751,610, Analysis A | 28 [25 to 31] | 27 [24 to 31]
  Week 24, n=624,529, Analysis B | 34 [30 to 38] | 32 [28 to 36]
  Week 36, n=751,610, Analysis A | 25 [22 to 29] | 30 [27 to 34]
  Week 36, n=482,461, Analysis B | 40 [35 to 44] | 40 [36 to 45]
  Week 48, n=751,610, Analysis A | 27 [24 to 30] | 35 [31 to 39]
  Week 48, n=454,433, Analysis B | 44 [40 to 49] | 49 [44 to 54]
  EOT, n=751,610, Analysis A | 34 [31 to 38] | 37 [33 to 41]
  EOT, n=571,496 Analysis B | 45 [41 to 49] | 46 [41 to 50]
  6 Months pt, n=751,610, Analysis A | 45 [41 to 49] | 51 [47 to 55]
  6 Months pt, n=542,475, Analysis B | 62 [58 to 66] | 65 [61 to 69]
  1 Year pt, n=751,610, Analysis A | 49 [45 to 53] | 51 [47 to 56]
  1 Year pt, n=492,432, Analysis B | 75 [71 to 78] | 73 [68 to 77]
  2 Year pt, n=751,610, Analysis A | 48 [45 to 52] | 53 [49 to 57]
  2 Year pt, n=461,419, Analysis B | 79 [75 to 82] | 77 [73 to 81]
  3 Year pt, n=751,610, Analysis A | 43 [40 to 47] | 49 [45 to 53]
  3 Year pt, n=405,366, Analysis B | 80 [76 to 84] | 82 [78 to 86]

11. Secondary Outcome: Alanine Transaminase Ratio Over Time by Hepatitis B Virus e Antigen Status
Description: ALT ratio was calculated as serum ALT, divided by the upper limit of the normal range.
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Ratio
  At Week 12, n=767, 807 | 2.07 (2.02) | 2.14 (2.07)
  At Week 24, n=702,770 | 1.92 (2.69) | 1.69 (1.32)
  At Week 36, n=542, 660 | 1.59 (1.57) | 1.42 (1.16)
  At Week 48, n=514,611 | 1.39 (1.13) | 1.23 (0.97)
  At EOT, n=645, 703 | 1.59 (2.34) | 1.38 (1.53)
  At 6 months post-trt, n=616, 673 | 1.19 (1.29) | 1.08 (1.48)
  At 1 year pt, n=551, 611 | 0.95 (0.98) | 0.96 (1.09)
  At 2 years pt, n=521, 594 | 0.86 (0.89) | 0.81 (0.65)
  At 3 years pt, n= 450, 519 | 0.83 (1.28) | 0.79 (0.88)

12. Secondary Outcome: Number of Participants With Chronic Hepatitis B - Associated Clinical Endpoints- Liver Transplantation, Hepatocellular Carcinoma, and Liver Decompensation
Description: Number of clinical endpoints associated with CHB reported in the medical record, where data available, are reported. The clinical endpoints included liver transplantation, hepatocellular carcinoma, liver decompensation, development of cirrhosis (in patients without cirrhosis at baseline).
Time Frame: Up to 276 Weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Participants
  Liver Transplantation, Yes | 0 | 1
  Hepatocellular Carcinoma, Yes | 4 | 7
  Liver Decompensation, Yes | 7 | 2

13. Secondary Outcome: Number of Participants With Chronic Hepatitis B Associated Clinical Endpoints- Liver Cirrhosis
Description: Number of participants with clinical endpoints associated with CHB captured in the medical record, where data available, are reported. The clinical endpoints included development of cirrhosis (in participants without cirrhosis at baseline). The liver cirrhosis assessments were summarized from Week 12 to 3 years post-treatment.
Time Frame: Up to 276 Weeks
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 844 | 872
Participants
  At Week 12, No Cirrhosis, n=73,89 | 59 | 82
  At Week 12, Transition To Cirrhosis, n=73,89 | 11 | 4
  At Week 12, Cirrhosis, n=73,89 | 3 | 3
  At Week 24, No Cirrhosis, n=73,94 | 58 | 77
  At Week 24, Transition To Cirrhosis, n=73,94 | 8 | 9
  At Week 24, Cirrhosis, n=73,94 | 7 | 8
  At Week 36, No Cirrhosis, n=36,67 | 30 | 58
  At Week 36, Transition To Cirrhosis, n=36,67 | 5 | 3
  At Week 36, Cirrhosis, n=36,67 | 1 | 6
  At Week 48, No Cirrhosis, n=44,80 | 35 | 66
  At Week 48, Transition To Cirrhosis, n=44,80 | 6 | 6
  At Week 48, Cirrhosis, n=44,80 | 3 | 8
  At 6 months, No Cirrhosis, n=116,158 | 102 | 134
  At 6 months, Transition To Cirrhosis, n=116,158 | 8 | 10
  At 6 months, Cirrhosis, n=116,158 | 6 | 14
  At 1 Year, No Cirrhosis, n=135,170 | 116 | 148
  At 1 Year, Transition To Cirrhosis, n=135,170 | 9 | 10
  At 1 Year, Cirrhosis, n=135,170 | 10 | 12
  At 2 Year, No Cirrhosis, n=132,175 | 121 | 153
  At 2 Year, Transition To Cirrhosis, n=132,175 | 7 | 14
  At 2 Year, Cirrhosis, n=132,175 | 4 | 8
  At 3 Years, No Cirrhosis, n=115,133 | 101 | 113
  At 3 Years, Transition To Cirrhosis, n=115,133 | 8 | 11
  At 3 Years, Cirrhosis, n=115,133 | 6 | 9

14. Secondary Outcome: Number of Participants With Serious Adverse Drug Reactions
Description: A serious adverse drug reactions (SADR) is any untoward medical occurrence suspected to be medicinal product-related that at any dose: Results in death, is life-threatening, NOTE: The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe. Requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or Is a congenital anomaly/birth defect.
Time Frame: Up to 276 Weeks
Population: Safety population was defined to include participants with informed consent who received at least one dose of PEG IFN and had at least one post-baseline safety assessment (any assessment after baseline).
Measure: Number; unit: Participants
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown
Number analyzed (Participants) | 863 | 890 | 48
Participants | 18 | 22 | 0

15. Secondary Outcome: Number of Participants With Non-Serious Adverse Drug Reactions
Description: Non serious adverse drug reactions (NSADRs) are all noxious and unintended responses to a medicinal product related to any dose.
Time Frame: Up to 276 Weeks
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown
Number analyzed (Participants) | 863 | 890 | 48
Participants | 585 | 599 | 28

16. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An Adverse Events (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes.
Time Frame: Up to 276 Weeks
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown
Number analyzed (Participants) | 863 | 890 | 48
Participants
  At Least One Adverse Event | 618 | 646 | 30
  At Least One Serious Adverse Event | 47 | 63 | 2

17. Secondary Outcome: Number of Deaths During Observation Period
Description: The clinical endpoint of deaths due to any cause during observation period is presented.
Time Frame: Up to 276 Weeks
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown
Number analyzed (Participants) | 863 | 890 | 48
Participants | 3 | 9 | 0

ADVERSE EVENTS:
Time Frame: Up to 276 Weeks
Description: Adverse Event (AE) is untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is with any of the following outcomes: Death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity; congenital anomaly.
Arm/Group | HBeAg Positive | HBeAg Negative | HBeAg Status Unknown
Serious Adverse Events (participants affected / at risk) | 47/863 | 63/890 | 2/48
Other Adverse Events (participants affected / at risk) | 522/863 | 562/890 | 30/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBeAg Positive (N=863) | HBeAg Negative (N=890) | HBeAg Status Unknown (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0
Dermoid Cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0
Basedow's Disease (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 2 | 0 | 0
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 0
Chest Pain (General disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatorenal Syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 3 | 2 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 3 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Cholangitis Infective (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 1 | 0
HIV Infection (Infections and infestations) | 0 | 1 | 0
Malaria (Infections and infestations) | 1 | 0 | 0
Meningitis Viral (Infections and infestations) | 0 | 2 | 0
Peritonitis Bacterial (Infections and infestations) | 0 | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia Haemophilus (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Tularaemia (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Open Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 2 | 0
Alpha 1 Foetoprotein Increased (Investigations) | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0
Thyroid Function Test Abnormal (Investigations) | 0 | 1 | 0
Transaminases Increased (Investigations) | 2 | 3 | 0
Tumour Marker Increased (Investigations) | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Coma (Nervous system disorders) | 0 | 1 | 0
Coma Hepatic (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0
Hepatic Encephalopathy (Nervous system disorders) | 2 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 1 | 0
Panic Attack (Psychiatric disorders) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hepatic Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic Stenosis (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HBeAg Positive (N=863) | HBeAg Negative (N=890) | HBeAg Status Unknown (N=48)
Anaemia (Blood and lymphatic system disorders) | 11 | 47 | 1
Leukopenia (Blood and lymphatic system disorders) | 55 | 125 | 6
Neutropenia (Blood and lymphatic system disorders) | 72 | 153 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 54 | 183 | 9
Nausea (Gastrointestinal disorders) | 33 | 28 | 4
Asthenia (General disorders) | 63 | 124 | 7
Fatigue (General disorders) | 89 | 93 | 3
Influenza Like Illness (General disorders) | 69 | 92 | 4
Pyrexia (General disorders) | 146 | 92 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 3 | 3 | 3
Weight Decreased (Investigations) | 58 | 76 | 7
White Blood Count Decreased (Investigations) | 73 | 18 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 48 | 35 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 81 | 74 | 2
Headache (Nervous system disorders) | 84 | 121 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 113 | 67 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 41 | 51 | 4

LIMITATIONS AND CAVEATS:
The study treatment was not harmonized as per local standard of care and possibly lead to country effects. Generalization of results was hampered by missing values. However, efficacy analyses endeavored to allow it by ITT and "as observed" approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.